CLINICAL TRIAL: NCT00289952
Title: Use of Valproic Acid to Purge HIV From Resting CD4+ Memory Cells/ A Proof-of-concept Study
Brief Title: Valproic Acid and Its Effects on HIV Latent Reservoirs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jean-Pierre Routy (Other)
Collaborators: Canadian Foundation for AIDS Research (CANFAR) (Other); CIHR Canadian HIV Trials Network (Network)
Responsible Party: Sponsor-Investigator, Jean-Pierre Routy, Dr Jean-Pierre Routy, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BMB#05-018 (CTN-205)
Record Dates: First submitted 2006-02-08; First posted 2006-02-10 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: HIV Infections
Keywords: HIV infections; Histone deacetylase Inhibitor; HIV Reservoirs; Peripheral Blood Mononuclear Cells; Valproic Acid; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Valproic Acid; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): HAART + valproic acid for 16 weeks followed by HAART alone for 32 weeks.
  Interventions: Drug: Valproic Acid; Drug: HAART
- Group 2 (Experimental): HAART alone for 16 weeks followed by HAART + valproic acid for 32 weeks.
  Interventions: Drug: Valproic Acid; Drug: HAART

INTERVENTIONS:
Drug: Valproic Acid — Oral valproic acid twice daily for 16 or 32 weeks. Dosage varies based on plasma levels.
Drug: HAART — As per standard of care.

SUMMARY:
The purpose of this study is to examine whether the co-administration of valproic acid (Epival®), with highly active antiretroviral therapy (HAART) can reduce the size of HIV latent reservoirs in infected CD4 cells.

DETAILED DESCRIPTION:
Participants must be on HAART with a suppressed viral load (< 50 copies/ml) for at least the previous 12 months. They will be randomly assigned to one of two groups, one group will start the valproic acid right away at week 1 for 16 weeks, and the other group will wait until week 17 to add valproic acid to their treatment for 32 weeks. Subjects will be followed every four weeks for one year and evaluated by a variety of assays, all carried out using well-established methods, to assess the main outcome defined by changes in HIV reservoir size measured by the mean frequency of resting CD4 memory cells carrying HIV proviral DNA.

ELIGIBILITY:
Inclusion Criteria:

Documented HIV seropositive infection by Western Blot, EIA assays or viral load.

* Aged 18 years old or older.
* Viral load <50 copies/ml for at least the previous 12 months.
* Circulating CD4+ cell count ³ 200 cells/ml.
* Taking HAART.
* Vital signs, physical examination and laboratory results do not exhibit evidence of diseases such as advanced cirrhosis and advanced liver disease (ALT or AST > 5 x upper limit of normal value).
* Karnofsky performance status 80%.
* Subject does not require and agrees not to take, for the duration of the study, any medication that is contraindicated with VPA.
* Willing and able to give informed consent.
* All participants will agree to abstinence or to used effective methods of contraception while on the study.

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Psychiatric or cognitive disturbance or illness that could preclude compliance with the study.
* Current use or use within four weeks prior to the baseline visit, of cytotoxic agents, systemic corticosteroids or any immunomodulatory agents such as intravenous immunoglobulin, or hydroxyurea.
* HIV vaccine within six months of screening visit
* Allergic reaction to VPA.
* Active intravenous drug users.
* History of bleeding disorders.
* Unstable or treated hypertension.
* Past-history of pancreatitis or chronic liver disease (ALT or AST > 5 x upper limit of normal value). However subject co-infected with hepatitis B or C can participate if ALT or AST is < 5 x upper limit of normal value.
* Renal failure (creatinine > 2 x upper limit of normal value).
* Ammonemia (> 2x upper limit of normal value).
* Taking Zidovudine (AZT), or combination of drugs containing AZT like Combivir or Trizivir. However this subject will be asked to switch to another NRTI,at least two weeks prior to Valproic Acid initiation, to become eligible.
* Taking on daily basis: phenytoin, carbamazepine, phenobarbital, warfarin or aspirin.
* Subject has any of the following abnormal laboratory results Hemoglobin < 100 g/L. Absolute neutrophil count < 0.75 x 10 9 cells/L. Platelet count < 50 x 10 9 cells/L.
* Subject suffering from urea cycle disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To assess the effect of VPA on HIV reservoirs measured by the frequency of resting CD4+ memory cells carrying HIV proviral DNA in peripheral blood of chronically HIV-infected subjects. | 16 or 32 weeks

SECONDARY OUTCOMES:
To assess the clinical and biological tolerance of VPA in chronically HIV-infected patients with undetectable viral load. | 16 or 32 weeks
To explore the changes in CD4/CD8 ratio, as the size of reservoir is thought to be inversely correlated with the frequency of resting CD4+ memory cells carrying HIV proviral DNA. | 48 weeks
To explore the frequency of CD4+ memory cell subsets (Tcm, Tpm and Tem) carrying HIV proviral DNA. | 48 weeks
To explore level of T-cell activation after VPA intervention. | 48 weeks
To assess levels of certain cytokines and chemokines, which are involved in T-cell proliferation and differentiation. | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Routy, MD, Principal Investigator — Royal-Victoria Hospital/McGill University Health Centre
Locations (6):
- Canada (6):
  - BC St-Paul's Hospital/Immunodeficiency Clinic, Vancouver, British Columbia
  - Ottawa Health Research Institute/Immunodeficiency Clinic, Ottawa, Ontario
  - Actuel Medical Clinic, Montreal, Quebec
  - Quartier Latin Medical Clinic, Montreal, Quebec
  - Montreal Chest Institute/Immunodeficiency Clinic, Montreal, Quebec
  - CHUL Ste-Foy, Ste-Foy, Quebec

REFERENCES:
- [Derived] Routy JP, Angel JB, Spaans JN, Trottier B, Rouleau D, Baril JG, Harris M, Trottier S, Singer J, Chomont N, Sekaly RP, Tremblay CL. Design and implementation of a randomized crossover study of valproic acid and antiretroviral therapy to reduce the HIV reservoir. HIV Clin Trials. 2012 Nov-Dec;13(6):301-7. doi: 10.1310/hct1306-301. PMID 23195668
- [Derived] Routy JP, Tremblay CL, Angel JB, Trottier B, Rouleau D, Baril JG, Harris M, Trottier S, Singer J, Chomont N, Sekaly RP, Boulassel MR. Valproic acid in association with highly active antiretroviral therapy for reducing systemic HIV-1 reservoirs: results from a multicentre randomized clinical study. HIV Med. 2012 May;13(5):291-6. doi: 10.1111/j.1468-1293.2011.00975.x. Epub 2012 Jan 26. PMID 22276680